CLINICAL TRIAL: NCT03699059
Title: A Study to Assess the Acceptability of an Online Weight Prevention Programme for New Kidney Transplant Recipients- The WEight Management in Renal Transplant Online Study (ExeRTiOn)
Brief Title: The wEight Management in Renal Transplant Online Study (ExeRTiOn)
Acronym: ExeRTiOn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Kidney Research U.K. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCH-EXERTION STUDY; 241928 (Other: IRAS project ID); KCH18-085 (Other: Sponsor site reference number (King's College Hospital))
Record Dates: First submitted 2018-08-08; First posted 2018-10-09 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Kidney Transplant; Complications; Obesity; Physical Activity; Weight Gain; Health Behavior
Keywords: Kidney transplant; Weight gain; Physical activity; Weight management
MeSH Terms: conditions — Obesity; Motor Activity; Weight Gain; Health Behavior | interventions — Physical Exertion

STUDY DESIGN:
Intervention Model Description: A small study creating a kidney transplant specific online weight gain prevention tool with qualitative data from 15 participants (5 transplant MDT members and 10 kidney transplant recipients)
Masking Description: No blinding. Purposive sampling of the 15 subjects- 5 HCP, 10 kidney transplant patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Care Professionals (Other): A purposeful sample of 5 HCP's from the transplant team will test the online intervention and be interviewed using qualitative methods. This data will be analysed and used to plan a second study (feasibility RCT).
  Interventions: Other: ExeRTiOn
- Kidney Transplant Patients (Other): A purposeful sample of 10 kidney transplant patients will test the online intervention and be interviewed using qualitative methods. This data will be analysed and used to plan a second study (feasibility RCT).
  Interventions: Other: ExeRTiOn

INTERVENTIONS:
Other: ExeRTiOn — REHAB-online is an online weight gain prevention tool comprising of physical activity advice, dietetic advice, self-monitoring and tracking and behavioural change techniques. This resource is specific to kidney transplant patients and has been created by the research steering group including patient representation. During this study participants (both HCPs and patients) will have a one-off study visit to test and evaluate the online intervention.

SUMMARY:
The primary aim of this project is to create an online weight management tool (Physical activity, weight management and cognitive behavioral therapy) to prevent significant weight gain following kidney transplantation. Designing the online interactive weight management resource for kidney transplant patients will involve patient and health care professional input through Qualitative methodology such as 'Think-Aloud' interviews and one-to-one semi-structured interviews. This online resource will be called "exertion" and will be created by the research team, with technical support from the Software Company (SPIKA).

Results from this study will refine the resource, and lead to a study application for a randomized controlled feasibility trial where we plan to test the "exertion" online application. Therefore this project has potential to influence clinical practice for kidney transplant recipients. It will allow patients, who may not have routine access to physio or dietetic input to address weight gain with support. A study flow chart summarizing the project can be found below.

DETAILED DESCRIPTION:
This study is a qualitative study and intervention planning study to create and refine an online resource for weight management in new kidney transplant (KTx) recipients, which will be named "exertion".

Objectives and hypothesis:

The aim of this qualitative study is to use qualitative methods to create and refine a weight management, exercise/ physical activity online resource for patients with kidney transplant recipients.

This study involves data collection via:

* Think-aloud interviews- 5 KTx patients and 2 Health Care Professionals (HCP) working in the transplant team will have recorded think aloud interviews using the resources. Other participants will be exposed to the resource during a routine lab session.
* Semi-structured interviews of transplant HCP's and KTx recipients.
* Demographic data including age, gender, occupation, smoking history, medical history, medication lists and baseline body weight (kg).
* Website/ resource log in data
* Field notes and observations from Think Aloud interviews, lab sessions and semi-structured interviews

The investigators aim to recruit 10 new kidney transplant recipients and 5 transplant health care professionals to explore the following themes through 'Think-Aloud' interviews:

* The functionality of the "exertion" online resource for KTx recipients
* The functionality of the "exertion" online resource from a HCP perspective
* KTx participants interpretation of the "exertion" modules and resource as a whole
* HCP participants interpretation of the "exertion" modules and resource as a whole
* Thought processes involved to use the "exertion" application
* Recommendations from participants
* Likes/dislikes
* Barriers/ easier to use sections
* Highlight individual differences in the use of the "exertion" resource

The investigators aim to explore the following themes through semi-structured individual interviews:

* What components of the online resource (exertion) are helpful/ unhelpful from a kidney transplant perspective?
* What components of the online resource are helpful/unhelpful from a kidney transplant HCP perspective?
* Are there any difficulties/ barriers participating in the study?
* And are they what were expected or different?
* Patients experiences and learning using the online application, and when the changes were noticed
* Anything missing/ they would recommend adding to the application

Statistical Analysis:

Baseline demographics of the participants will be described using summary statistics. Continuous variables will be summarized using the mean and standard deviation (SD) if approximately normally distributed. Continuous variables that are not normally distributed will be summarized using the median and IQR.

Qualitative analysis: Data will be collected through in-depth feedback about the online intervention materials; field notes, individual interviews and 'Think-aloud' interviews. 'Think-aloud' interviews will be used to elicit participants' reactions to sessions of the online intervention; participants will be observed and asked to comment aloud on reactions to every aspect of the different sessions. Semi-structured interviews will explore participants' overall impressions of the online intervention. These qualitative techniques will allow for themes and sub-themes to emerge. The website will be designed to record user entries, and observational field notes about participants' use of the intervention will also be collected. Individual interviews will be transcribed verbatim and analysed using an inductive thematic analysis approach (17), informed by techniques of grounded theory (15), including line-by-line open coding grounded in data and constant comparison of all instances of codes. Deviant case codes will be employed to ensure that perspectives that diverge from dominant trends are not overlooked.

ELIGIBILITY:
Eligibility criteria for the Kidney Transplant Participants (n=10)

Inclusion Criteria:

* adult patients (18years+)
* Male or female
* Written informed consent
* < 3 months post kidney transplant
* access to internet connected computer, smart-phone or tablet
* A Body Mass Index (BMI) greater than or equal to 18.5 (healthy range)

Exclusion Criteria:

* pregnancy
* Unstable medical conditions such as; angina, uncontrolled hypertension or diabetes, congestive cardiac failure, active myocarditis/ pericarditis, cardiac arrhythmia, co-morbid catabolic conditions, psychiatric illness.
* Participated in a structured exercise or physical activity intervention in the last three months.
* BMI of less than 18.5 (classified as underweight)
* significant cognitive impairment preventing them from engaging with online interactive material

Eligibility criteria for the Transplant Health Care Professionals (n=5)

Inclusion criteria:

* A nephrologist, kidney doctor, nurse or member of the multi-disciplinary team who actively work with kidney transplant patients at King's College Hospital
* Adult above 18 years of age
* Able to provide written consent
* Access to Internet connected computer, smart-phone or tablet.

Exclusion criteria:

* Pregnancy
* Unstable medical conditions such as angina, uncontrolled hypertension or diabetes, congestive cardiac failure, active myocarditis, cardiac arrhythmia, co-morbid catabolic condition, psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Patient experience and learning using the "ExeRTiOn" online resource | day 1
  Patient experience and learning using the "ExeRTiOn" online resource determined by qualitative interview

SECONDARY OUTCOMES:
Transplant health care professional experience and knowledge reviewing the online resource | day 1
  Transplant health care professional experience and knowledge reviewing the online resource determined by qualitative interview
Any difficulties/ barriers to participating in the study | day 1
  Any difficulties/ barriers to participating in the study determined by a qualitative interivew
Any difficulties/ barriers to using the "ExeRTiOn" resource | day 1
  Any difficulties/ barriers to using the "ExeRTiOn" resource determined by a qualitative interview
Components of the "ExeRTiOn" resource that are helpful/ unhelpful | day 1
  Transplant health care professional experience and knowledge reviewing the online resource determined by qualitative interview
Weakness of the "ExeRTiOn" resource | day 1
  Weakness of the "ExeRTiOn" resource determined by a qualitative interview
Strengths of the "ExeRTiOn" resource | day 1
  Strengths of the "ExeRTiOn" resource determined by a qualitative interview
feasibility and use of the ExeRTiOn resource | day 1
  log in time for the study visit and time using the resource will be recorded by the online resource
feasibility outcome (adherence) | day 1
  adherence to study visits
height | day 1
  measured in centimeters
weight | day 1
  measured in kilograms
Body mass index (BMI) | day 1
  weight and height will be combined to report BMI in kg/m2
descriptive data | day 1
  descriptive data including gender, date of transplant and age

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Castle, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The research team plan to make de-identified participant data available as supplementary material to an online publication
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: within 6-12 months of study completion
Access Criteria: data will be available as supplementary material through online publication. For example Plos one.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT03699059/Prot_SAP_000.pdf